CLINICAL TRIAL: NCT04256538
Title: Identify Specific PBMC miRNAs as Biomarkers for IBD
Brief Title: Identify Specific Peripheral Blood Mononuclear Cell (PBMC) MiRNA as Biomarkers for Inflammatory Bowel Disease (IBD)
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHZJU2019-189
Record Dates: First submitted 2020-01-16; First posted 2020-02-05 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Crohn's Disease Group: Patients are diagnosed as Crohn's disease and have no history of colectomy.
- Ulcerative Colitis Group: Patients are diagnosed as ulcerative colitis and have no history of colectomy.
- Healthy Control Group: Individuals that have no past medical history.

SUMMARY:
To find high sensitivity and specificity biomarkers to better diagnose and monitor progression of inflammatory bowel disease (IBD). In this study, we try to find miRNAs that can used to diagnose or monitor progression of IBD by exploring differential expression of miRNAs in peripheral blood mononuclear cells (PBMCs) from Crohn's disease, ulcerative colitis and healthy controls. And we further validate these miRNAs in a larger population to assess their function as biomarkers.

DETAILED DESCRIPTION:
Incidence of inflammatory bowel disease (IBD) has been rising in the past decades. However, diagnosis and differential diagnosis of IBD still lack gold standard. To diagnose IBD, physicians need to combine clinical manifestation, lab results, image examination, endoscopy examination and pathology. After diagnosis, patients still need to monitor their disease progression. The most accurate way is to do endoscopy examination, however, endoscopy examination is an invasive, expensive and uncomfortable procedure. At present, C-reactive protein (CRP), erythrocyte sedimentation rate (ESR) and fecal calprotectin are used as main noninvasive biomarkers to monitor progression routinely. But their specificities are still unsatisfactory. So, it's urgent to find high sensitivity and specificity biomarkers to better diagnose and monitor progression of IBD. In this study, we try to find miRNAs that can used to diagnose or monitor progression of IBD by exploring differential expression of miRNAs in peripheral blood mononuclear cells (PBMCs) from Crohn's disease, ulcerative colitis and healthy controls. And we further validate these miRNAs in a larger population to assess their function as biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as Crohn's disease (CD) or ulcerative colitis (UC) according to World Health Organization (WHO) criteria
* Vital signs are stable

Exclusion Criteria:

* Refuse to sign consent
* Refuse to do examination to assess their disease progression
* CD patients only upper gastrointestinal tract (GI) is involved (L4)
* Had colectomy or in artificial opening status
* Have other autoimmune comorbidity
* Had severe infection within a week
* Had surgery within a month
* Have malignant tumor
* Pregnancy or lactation

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 14-75 years old, diagnosed as CD or UC according to WHO criteria, are recruited at specialist IBD clinic. They are excluded if upper GI is the only involved part, had colectomy or in artificial opening status or have other autoimmune comorbidity.
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index (CDAI) | 2 months
  Crohn's Disease Activity Index (CDAI) has been developed to assess whether or not the pathology of Crohn's disease is progressing.
  The index is the sum of 8 components, to each of which is assigned a specific weight. <150 suggests remission, 151-219 suggests mild activity, 220-450 suggests moderate activity, >450 suggests severe activity
Mayo Score | 2 months
  The full Mayo Score evaluates ulcerative colitis stage, based on four parameters: stool frequency, rectal bleeding, endoscopic evaluation and Physician's global assessment.
  Each parameter of the score ranges from zero (normal or inactive disease) to 3 (severe activity).
  0-2 suggests remission, 3-5 suggests mild activity,6-10 suggests moderate activity, >10 suggests severe activity

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China